CLINICAL TRIAL: NCT01855074
Title: Evaluation of Efficacy and Safety of Risperidone in Long-acting Microspheres in Patients With Schizophrenia, Schizophreniform or Schizoaffective Disorders Diagnosed According to the DSM-IV Criteria, After Switching Treatment With Any Antipsychotic Therapy With Long-acting Microspheres of Risperidone
Brief Title: An Efficacy and Safety Study of Risperidone Long-Acting Microspheres in Participants With Schizophrenia, Schizophreniform or Schizoaffective Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR014845; RISSCH4186
Record Dates: First submitted 2013-03-22; First posted 2013-05-16 (Estimated); Results first posted 2013-07-25 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Schizophrenia; Schizophreniform Disorder; Schizoaffective Disorder
Keywords: Schizophrenia; Schizophreniform Disorder; Schizoaffective Disorder; Risperidone; Risperdal consta
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Risperidone (Experimental): Risperidone 25 milligram (mg) will be given as intramuscular injection for every 2 weeks up to 6 months. Participants with persistent symptoms and/or requiring higher doses of antipsychotics will be administered higher doses of risperidone. Doses will be adjusted as per Investigator's discretion.
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Risperidone — Risperidone 25 milligram (mg) will be given as intramuscular injection for every 2 weeks up to 6 months. Participants with persistent symptoms and/or requiring higher doses of antipsychotics will be administered higher doses of risperidone. Doses will be adjusted as per Investigator's discretion.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of long acting injectable microspheres of risperidone in participants with schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self), schizophreniform or schizoaffective disorders (disorders in which there is a loss of ego boundaries or a gross impairment in reality testing with delusions or prominent hallucinations).

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), longitudinal (participants are followed over time with continuous or repeated monitoring of risk factors or health-outcomes), non-randomized (a clinical trial in which the participants are not assigned by chance to different treatment groups), single-center study to evaluate the efficacy and safety of long acting microspheres of risperidone in adult participants with schizophrenia, schizophreniform or schizoaffective disorders. The duration of this study will be 12 months and duration of treatment will be 6 months. The study will include 4 visits: Baseline, and 3 follow-up visits including Week 4, 12 and 26. All eligible participants will be treated with risperidone 25 milligram (mg) intramuscular injection (injection of a substance into a muscle) for every two weeks up to 6 months. Participants with persistent symptoms and/or requiring higher doses of antipsychotics (agents that control agitated psychotic behavior, alleviate acute psychotic states, reduce psychotic symptoms, and exert a quieting effect) will be initiated with higher doses of risperidone. Doses will be adjusted according to the response of the treatment. Efficacy and safety of the participants will be primarily evaluated by Positive and Negative Syndromes Scale (PANSS) and Extrapyramidal Symptom Rating Scale (ESRS), respectively. Participants' quality of life and safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatically stable participants defined as a) participants with treatment on outpatient and inpatient basis for at least 4 weeks before entering the study, and b) Positive and Negative Syndrome Scale (PANSS) Positive Subscale Score less than or equal to (<= ) 3 (1-7), including conceptual disorganization, suspicion, hallucinatory conduct and delirium (state of violent mental agitation)
* Participants under antipsychotic treatment with extrapyramidal symptoms, persistent negative symptoms or lack of adherence defined as irregular administration of medication in the last 2 weeks
* Participants who have given their informed consent in writing, or at least, by their family member or personal representative

Exclusion Criteria:

* Participants taking first antipsychotic treatment in his/her life
* Participants with any other psychotic disorder different to the previously mentioned in the inclusion criteria
* Pregnant or nursing women
* History of neuroleptic malignant syndrome (potentially fatal syndrome associated primarily with the use of antipsychotic drugs and clinical features include diffuse muscle rigidity, tremor, high fever) or current symptoms of tardive dyskinesia (a neurological disorder characterized by involuntary movements of the face and jaw)
* Participants with known intolerance or lack of response to risperidone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd. Clinical trial, Study Director — Janssen-Cilag Ltd.

RESULTS

PARTICIPANT FLOW:
Groups:
- Risperidone: Risperidone 25 milligram (mg) was administered as intramuscular injection (injection of a substance into a muscle) every 2 weeks up to 6 months
Period: Overall Study
Arm/Group | Risperidone
Started | 80
Treated | 79
Completed | 66
Not Completed | 14
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 8
Not completed — Started but not treated | 1

BASELINE CHARACTERISTICS:
Arm/Group | Risperidone
Number analyzed (Participants) | 79
Age Continuous [Mean (Standard Deviation); unit: Years] — Safety set (SS) population (N=79) included all participants who received at least 1 dose of study drug.
  Years | 43.0 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Safety set (SS) population (N=79) included all participants who received at least 1 dose of study drug.
  Participants
    Female | 32
    Male | 47

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Week 26
Description: The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 to 210, higher scores indicate worsening. Change at Week 26 score is calculated as Baseline score minus Week 26 score.
Time Frame: Baseline and Week 26
Population: The Intent-to-treat (ITT) population included all the participants who received at least 1 dose of study medication and had at least 1 follow-up visit. Here 'n' signifies number of participants evaluable for this outcome measure at specific time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Risperidone
Number analyzed (Participants) | 78
Units on a scale
  Baseline (n=78) | 68.9 (15.8)
  Change at Week 26 (n=66) | 28.1 (17.1)

2. Secondary Outcome: Clinical Global Impressions (CGI) - Disease Severity Score
Description: The CGI rating scale is a 7-point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants", higher scores indicate worsening.
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Risperidone
Number analyzed (Participants) | 78
Units on a scale
  Baseline (n=78) | 4.2 (4.0)
  Week 26 (n=66) | 2.9 (3.0)

3. Secondary Outcome: Short Form-36 (SF-36) - Quality of Life Score
Description: The SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: vitality, physical function, social function, physical role, emotional role, bodily pain, general health, mental health. Each item is scored on a scale ranging from 0-100 (100=highest level of functioning).
Time Frame: Baseline and Week 26
Population: The ITT population included all the participants who received at least 1 dose of study medication and had at least 1 follow-up visit. Here, 'n' signifies number of participants evaluable for this outcome measure at specific time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Risperidone
Number analyzed (Participants) | 78
Units on a scale
  Baseline; Physical function (n=78) | 78.3 (21.7)
  Week 26; Physical function (n=66) | 90.5 (13.8)
  Baseline; Physical role (n=78) | 41.0 (46.5)
  Week 26; Physical role (n=66) | 75.4 (41.0)
  Baseline; Body pain (n=78) | 86.2 (19.8)
  Week 26; Body pain (n=66) | 94.7 (11.8)
  Baseline; General health (n=78) | 51.7 (18.3)
  Week 26; General health (n=66) | 67.8 (12.0)
  Baseline; Vitality (n=78) | 51.7 (16.8)
  Week 26; Vitality (n=66) | 58.6 (11.5)
  Baseline; Social function (n=78) | 49.0 (20.4)
  Week 26; Social function (n=66) | 74.1 (18.1)
  Baseline; Emotional role (n=78) | 32.1 (46.0)
  Week 26; Emotional role (n=66) | 73.2 (42.3)
  Baseline; Mental health (n=78) | 50.7 (13.8)
  Week 26; Mental health (n=66) | 59.9 (12.8)

4. Secondary Outcome: Global Assessment of Functioning (GAF) Score
Description: The GAF is a 100-point tool to measure overall psychological, social and occupational functioning of adults. The higher score range (91 to 100) refers to a superior functioning in a wide range of activities, and absence of symptoms. The lower score range (1 to 10) refers to persistent danger of severely hurting self or others; or persistent inability to maintain minimum personal hygiene; or serious suicidal act with clear expectation of death.
Time Frame: Baseline and Week 26
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Risperidone
Number analyzed (Participants) | 78
Units on a scale
  Baseline (n=78) | 56.5 (14.2)
  Week 26 (n=66) | 69.4 (11.7)

5. Secondary Outcome: Patient Satisfaction With Treatment
Description: Participants' were assessed for their satisfaction with the current antipsychotic treatment on a 5-point scale/questionnaire: very good, good, reasonable, moderate or poor.
Time Frame: Baseline and Week 26
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Risperidone
Number analyzed (Participants) | 78
Participants
  Baseline; Very good (n=78) | 2
  Week 26; Very good (n=66) | 16
  Baseline; Good (n=78) | 13
  Week 26; Good (n=66) | 40
  Baseline; Moderate (n=78) | 42
  Week 26; Moderate (n=66) | 10
  Baseline; Poor (n=78) | 19
  Baseline; Very poor (n=78) | 1
  Baseline; No available (n=78) | 1

6. Secondary Outcome: Extrapyramidal Symptom Rating Scale (ESRS) Score
Description: An ESRS scale is used to assess the extrapyramidal symptoms attributable to antipsychotics. It consists of 8 items to assess individual symptoms and each item is assessed from 0 (none, absent) to 4 (severe). The total score is the sum of the 8 item scores, for a total range of 0 (normal) to 32 severe). The items for the assessment of individual symptoms are classified into 4 categories of parkinsonism, akathisia, dystonia and dyskinesia.
Time Frame: Baseline and Week 26
Population: Safety set (SS) population (N=79) included all participants who received at least 1 dose of study drug. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Risperidone
Number analyzed (Participants) | 78
Units on a scale
  Baseline | 12.9 (9.6)
  Week 26 | 9.2 (5.1)

ADVERSE EVENTS:
Description: Safety set (SS) population (N=79) included all participants who received at least 1 dose of study drug.
Arm/Group | Risperidone
Serious Adverse Events (participants affected / at risk) | 1/79
Other Adverse Events (participants affected / at risk) | 1/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Risperidone (N=79)
Psychotic disorder (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Risperidone (N=79)
Extrapyramidal disorder (Nervous system disorders) | 1

LIMITATIONS AND CAVEATS:
The planned sample size was not reached and a high dropout rate of participants was observed. Due to the high number of protocol violations, analysis was performed as intention-to-treat instead of per protocol as was planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the information generated through services from the Principal Investigator (PI), the Sponsor has the rights to publish the data without previous consent from the PI.

The PI must not publish completely or partially any results from the study, without previous authorization from the Sponsor.